CLINICAL TRIAL: NCT03986983
Title: Effect of Shockwave Therapy Associated With an Aerobic Exercise Program on the Degree of Severity of Gynoid Lipodystrophy in Women: a Randomized Controlled Trial
Brief Title: Shockwave Therapy (SWT)
Acronym: SWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Investigator- Integrated Researcher, Center for Rehabilitation Research (CIR) School of Health of P.PORTO., Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AN-008
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Gynoid Lipodystrophy
Keywords: Gynoid Lipodystrophy; Shock Wave Therapy; Aerobic Exercise
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group of Aerobic exercise (Experimental): The participants perform the Aerobic exercise protocol - The entire protocol was monitored through the Polar® brand heart rate monitor and watch.
  Interventions: Other: Aerobic exercise
- Experimental group of Shockwave therapy and Aerobic Exercise (Experimental): The participants do the Shockwave therapy protocol - The shockwave therapy protocol was performed in the prone position.
  In addition, the participants also perform the Aerobic exercise protocol - The entire protocol was monitored through the Polar® brand heart rate monitor and watch.
  Interventions: Device: Shockwave therapy; Other: Aerobic exercise
- Control group (No Intervention): The participants do not perform any type of intervention.

INTERVENTIONS:
Device: Shockwave therapy — Shockwave therapy protocol - The shockwave therapy protocol was performed in the prone position. The application was radial shockwave with 3,5bar, 15Hz of frequency and 3000 impulses.
  Arms: Experimental group of Shockwave therapy and Aerobic Exercise
Other: Aerobic exercise — Aerobic exercise protocol - 30 minutes of aerobic moderate-intensity exercise (40% of reserve heart rate) using Karvonen´s formula, performed on a step.
  Arms: Experimental group of Aerobic exercise; Experimental group of Shockwave therapy and Aerobic Exercise

SUMMARY:
The purpose of the present study is to evaluate the effects of six sessions of aerobic exercise associated with shock waves therapy in the severity of gynoid lipodystrophy.

DETAILED DESCRIPTION:
The Gynoid Lipodystrophy (GL) is considered to be a subcutaneous tissue disorder that causes changes in visible skin topography in the form of protrusions and depressions, mainly located in the lower limbs and abdominal region. It is a non-inflammatory and degenerative condition whose etiology has not been fully elucidated until now, although it can be explained by varied theories: the hormonal ,that is related to estrogen, the morphological one, based on alterations of the adipose tissue that is related to the interlobular septa of connective tissue that interconnects the subcutaneous adipose lobes, these septa are thin and have perpendicular projections, which favors the deposition of adipose tissue and its expansion to the surface of the dermis. The last one is about microcirculation deficits that can lead to intracellular edema and reduction of lymphatic drainage.

Shock wave therapy appears to be a safe and effective therapy to act in this disorder. It generates mechanical pressure waves in the tissues, promoting cavitation phenomena that produces lipolysis by destroying the cell membrane of adipocytes, increasing blood flow in the region, and stimulating lymphatic drainage.

On the other hand, there are studies that report that improvement in the appearance of GL is associated with a decrease in subcutaneous adipose tissue. Physiologically, aerobic physical exercise has the capacity to decrease body fat, taking into account that the oxidation reactions of fatty acids are enhanced, with moderate intensity exercise.

In this sense, it may be beneficial to associate Shockwave Therapy and Physical Exercise to reduce GL severity, so this study aims to analyze the effect of radial shock wave therapy in association with the performance of an aerobic exercise program, in female subjects, in the degree of GL severity in the gluteal region and ⅓ proximal posterior of the thighs.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a moderate and severe degree of cellulitis, according to an CSS, in the region of the buttocks and ⅓ proximal posterior of the thighs;

Exclusion Criteria:

* Unstable weight during the last 6 months, with a variation of less than or equal to 2 kg has been initiated;
* Hormonal treatment (contraceptive pill, intrauterine device, other) changed in the last 6 months;
* Participants with food restrictions;
* Pregnant women or post childbirth during the last year;

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Change in the score of the Cellulite Severity Scale (CSS) | before the intervention program
  Verified by changes in the score of the CSS. The CSS is used to measure the severity of GL, this scale quantifies 5 variables such as the number of evident depressions, the depth of depressions , the morphological aspect of the skin surface, the degree of laxity, flaccidity, or sagging skin and the classification of GL using the scale of Nurnberger and Muller. Each variable can have a score of 0 to 3 and the final score is made by the total sum of these. The final score goes from 0 to 15 , which means that 0 to 5 is a mild degree of GL, 6 to 10 is moderate degree and 11 to 15 is considered a severe degree.

SECONDARY OUTCOMES:
Subcutaneous buttock tissue thickness | before the intervention program
  Verified by changes in the measurement of the subcutaneous adipose fold by ultrasonography (mm)
Changes in anthropometric measurements such as hip circumference, gluteal fold, and the proximal ⅓ of the thigh | before the intervention program
  Verified by changes in anthropometric measures such as hip circumference, gluteal fold, and the proximal ⅓ of the thigh before and after the intervention, evaluated using a tape measure (cm)
Change in the microcirculation of the treatment area | before the intervention program
  Verified by changes in the thermography (ºC)

CONTACTS AND LOCATIONS:
Locations (1):
- Andreia Noites, Porto, Portugal

REFERENCES:
- [Background] Adatto M, Adatto-Neilson R, Servant JJ, Vester J, Novak P, Krotz A. Controlled, randomized study evaluating the effects of treating cellulite with AWT/EPAT. J Cosmet Laser Ther. 2010 Aug;12(4):176-82. doi: 10.3109/14764172.2010.500392. PMID 20590369
- [Background] Adatto MA, Adatto-Neilson R, Novak P, Krotz A, Haller G. Body shaping with acoustic wave therapy AWT((R))/EPAT((R)): randomized, controlled study on 14 subjects. J Cosmet Laser Ther. 2011 Dec;13(6):291-6. doi: 10.3109/14764172.2011.630089. PMID 21981441
- [Background] Christ C, Brenke R, Sattler G, Siems W, Novak P, Daser A. Improvement in skin elasticity in the treatment of cellulite and connective tissue weakness by means of extracorporeal pulse activation therapy. Aesthet Surg J. 2008 Sep-Oct;28(5):538-44. doi: 10.1016/j.asj.2008.07.011. PMID 19083577
- [Background] Hexsel D, Camozzato FO, Silva AF, Siega C. Acoustic wave therapy for cellulite, body shaping and fat reduction. J Cosmet Laser Ther. 2017 Jun;19(3):165-173. doi: 10.1080/14764172.2016.1269928. Epub 2017 Feb 2. PMID 27997260
- [Background] Knobloch K, Joest B, Kramer R, Vogt PM. Cellulite and focused extracorporeal shockwave therapy for non-invasive body contouring: a randomized trial. Dermatol Ther (Heidelb). 2013 Dec;3(2):143-55. doi: 10.1007/s13555-013-0039-5. Epub 2013 Dec 3. PMID 24297647
- [Background] Modena DAO, da Silva CN, Grecco C, Guidi RM, Moreira RG, Coelho AA, Sant'Ana E, de Souza JR. Extracorporeal shockwave: mechanisms of action and physiological aspects for cellulite, body shaping, and localized fat-Systematic review. J Cosmet Laser Ther. 2017 Oct;19(6):314-319. doi: 10.1080/14764172.2017.1334928. Epub 2017 Jun 7. PMID 28590827
- [Background] Perez Atamoros FM, Alcala Perez D, Asz Sigall D, Avila Romay AA, Barba Gastelum JA, de la Pena Salcedo JA, Escalante Salgado PE, Gallardo Palacios GJ, Guerrero-Gonzalez GA, Morales De la Cerda R, Ponce Olivera RM, Rossano Soriano F, Solis Tinoco E, Welsh Hernandez EC. Evidence-based treatment for gynoid lipodystrophy: A review of the recent literature. J Cosmet Dermatol. 2018 Dec;17(6):977-983. doi: 10.1111/jocd.12555. Epub 2018 Apr 30. PMID 29707877